CLINICAL TRIAL: NCT02299362
Title: The Treatment of Progressive Early Onset Spinal Deformities: A Multi-Center Outcome Study
Acronym: GSSG
Status: Completed | Type: Observational
Sponsor: Growing Spine Study Group (Other)
Collaborators: Growing Spine Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB-08055C
Record Dates: First submitted 2014-11-18; First posted 2014-11-24 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Early Onset Scoliosis; Congenital Spinal Deformities; Infantile Idiopathic Scoliosis; Neuromuscular Spinal Deformity; Syndromic Spinal Deformity; Thoracic Insufficiency Syndrome
Keywords: Early Onset Scoliosis; EOS; Pulmonary function; Infantile Idiopathic Scoliosis; MCGR; Magnetically controlled growing rods; Growing rods; Growth friendly spine surgery; Cast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to examine the treatment, both surgical and non-surgical, of patients with any form of early onset scoliosis. Such treatment may include the use of growth friendly devices that are surgically or magnetically lengthened; or the use of serial body casting or bracing, or observation. Outcomes examined will be what can be seen physically on the patient and on x-ray, as well as parent perception of how the treatment effects their child with the use of a health-related quality of life (HRQOL) questionnaire.

DETAILED DESCRIPTION:
This multi-center study will evaluate the long-term clinical and radiographic outcomes of Early Onset Scoliosis (EOS) and other Early Onset Spinal and Chest Wall Deformities in a large population of patients.

The study will attempt to answer the following clinical questions:

1. How do clinical parameters (e.g. height, weight, pulmonary function, incidence of complications) differ between:

   1. Age groups
   2. Etiologic groups
   3. Treatment types including operative and non-operative methods
   4. Patients who receive definitive spinal fusion versus those who do not
2. How do radiographic parameters (e.g. curve size, spinal height, thoracic dimensions, sagittal profile, pelvic parameters, spinal balance) differ between:

   1. Age groups
   2. Etiologic groups
   3. Treatment types including operative and non-operative methods
   4. Patients who receive definitive spinal fusion versus those who do not
3. How does health-related quality of life (HRQOL), using the EOSQ-24 outcomes tool, differ between:

   1. Age groups
   2. Etiologic groups
   3. Treatment types including operative and non-operative methods
   4. Patients who receive definitive spinal fusion versus those who do not
4. What demographic, clinical, radiographic, and surgical factors contribute to the incidence of complications?
5. For patients with a particular diagnosis, age and/or treatment type, what are the clinical, radiographic and HRQOL changes before and after treatment?
6. What are the mechanisms that cause rod breakage in growing rod constructs? (This study question is a collaborative research study with the U.S. Food and Drug Administration).

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age and any diagnosis who undergo a growth-friendly surgical procedure, including but not limited to growing rods, VEPTR, Shilla, hybrid constructs, spinal tethering and staples
* Patients of any age and any diagnosis who undergo casting
* Patients of any diagnosis 10 years of age and younger who undergo spinal fusion of the thoracic and/or lumbar spine
* Patients of any diagnosis under 6 years of age with scoliosis curves of the thoracic and/or lumbar spine measuring > 25 degrees. Observed and braced patients included

Exclusion Criteria:

* Cervical spine anomalies alone will not be included
* Patient/family is unwilling to participate in the study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients receiving treatment at participating study sites who are eligible and agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 2602 (Actual)
Dates: Start 2008-10; Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Clinical and Radiographic | 18 years
  Evaluation of long-term clinical measures such as: BMI, Pulmonary functionality, incidence of complications; and radiographic outcomes (e.g. coronal spinal curvature, sagittal profile, spinal and thoracic growth, coronal and sagittal alignment.

SECONDARY OUTCOMES:
Patient based outcomes | 18 years
  Evaluation of the effect of treatment on patients and families by use of serial early-onset scoliosis questionnaire (EOSQ-24) scores during treatment. EOSQ covers the following domains: Child's Health Related Quality of Life (16 items), Family Impact (2 items) and Satisfaction (2 items).

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Sponseller, MD, MBA, Principal Investigator — Johns Hopkins Bloomberg Children's Center
Locations (27):
- United States (19):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Nemours/Alfred I. Dupont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Indiana University Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - C.S. Mott Childrens Hospital, Ann Arbor, Michigan
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - University of Rochester, Rochester, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Scottish Rite Hospital for Children, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hospital Sainte-Justine, Montreal, Quebec
- Cairo University, Giza, Egypt
- FOCOS Orthopaedic Hospital, Accra, Pantang West, Ghana
- Spain (2):
  - Hospital Unversitario La Paz, Madrid
  - Hospitales Unversitarios Virgen del Rocio, Seville
- Hacettepe University, Ankara, Turkey (Türkiye)
- Royal Orthopaedic Hospital, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data stored in the GSSG database will also be shared with 24 sites that comprise the Children's Spine Study Group (CSSG). The collaboration between GSSG and CSSG is solely for research purposes.
  Fully de-identified data from the GSSG database may be shared with key stakeholders including, but not limited to, medical device companies, professional societies, regulatory agencies, patients and surgeons to support endeavors that are aimed to improve the care of EOS patients. These data may be shared to support the following activities:
  1. Filings for medical device clearance by the U.S. Food and Drug Administration (FDA)
  2. Health care cost assessments
  3. Future clinical research studies on EOS

REFERENCES:
- See also: Growing Spine Foundation webpage — https://www.growingspine.org/research